CLINICAL TRIAL: NCT07240961
Title: Ultrasound-Guided Lumbal Erector Spinae Plane Block on Postoperative Pain Management After Total Hip Arthroplasty
Brief Title: Lumbal Erector Spinae Plane Block for Pain Management After Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, professor, University Tunis El Manar
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IMKO-CE 115/2024
Record Dates: First submitted 2025-05-01; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-05

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: hip arthroplasty; Lumbal Erector Spinae Plane Block; pain managment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hip arthroplasty with nerve block (Active Comparator): Lumbar ESP block performed after anesthesia induction. A low-frequency ultrasound probe will be placed longitudinally 2-3 cm lateral to the L4 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle (100 mm, 22G) will be inserted cranio-caudal direction and following confirmation of the correct position of the needle, between the erectorspinae muscle and the transverse process,30 ml of local anesthetic (0.25% bupivacaine/0.2% ropivacaine) will be administered for the block
  Interventions: Procedure: Lumbal Erector Spinae Plane Block
- hip arthroplasty with intravenous pain killers (Placebo Comparator): intravenous pain killers
  Interventions: Procedure: intravenous pain killers

INTERVENTIONS:
Procedure: Lumbal Erector Spinae Plane Block — Lumbar ESP block performed after anesthesia induction. A low-frequency ultrasound probe will be placed longitudinally 2-3 cm lateral to the L4 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle (100 mm, 22G) will be inserted cranio-caudal direction and following confirmation of the correct position of the needle, between the erectorspinae muscle and the transverse process,30 ml of local anesthetic (0.25% bupivacaine/0.2% ropivacaine) will be administered for the block.
  Arms: hip arthroplasty with nerve block
Procedure: intravenous pain killers — intravenous pain killers
  Arms: hip arthroplasty with intravenous pain killers

SUMMARY:
The Erector Spinae Plane (ESP) block or spinal erector block was first described in September 2016 by a Canadian team. It's a block that was initially used for the treatment of chronic thoracic neuropathic pain. The ESP block is one of the inter-fascicular blocks and it's an easy-to-perform technique.In the literature, it has been reported that Lumbar ESPB provides effective analgesia after a hip surgery.

The purpose of this prospective randomized study was to compare the analgesic effects of the ultrasound-guided lumbar Erector Spinae Plane block on postoperative pain management versus the multimodal analgesia after total hip arthroplasty.

DETAILED DESCRIPTION:
Patients aged more than 18 years, ASA I-III scheduled for primary total hip arthroplasty with lateral approach and under general anesthesia Patients were randomly assigned, into 1 of 2 groups, namely, group ESPBL and group Placebo, using sealed envelopes

* For ESPBL group: Lumbar ESP block performed after anesthesia induction. A low-frequency ultrasound probe will be placed longitudinally 2-3 cm lateral to the L4 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle (100 mm, 22G) will be inserted cranio-caudal direction and following confirmation of the correct position of the needle, between the erectorspinae muscle and the transverse process,30 ml of local anesthetic (0.25% bupivacaine/0.2% ropivacaine) will be administered for the block.
* For Placebo group: patients had multimodal analgesia without lumbar ESP block Patients will be transferred to continuous care unit for 24 hours.

Post-operative analgesia will include:

1. Paracetamol 1g IV every 8 hours for 1 day then oral paracetamol 1g every 8 hours for 4 weeks.
2. Diclofenac sodium(50mg) 1 tablet x 2 per day for 5 days.
3. PCA morphine (Patient Controlled Analgesia), as a rescue analgesia, programmed as: Bolus of 1mg/ refractory period of 10 min/ maximum dose set up at 10mg every 12h.

The primary outcome of the study is to compare postoperative opioids consumption in the first 24 postoperative hours.

Secondary endpoints:

Secondary outcomes are: intraoperative opioid consumption, postoperative pain scores, sitting position and adverse effects related to opioids.

ELIGIBILITY:
Inclusion Criteria:

* primary total hip arthroplasty with lateral approach and under general anesthesia .

Exclusion Criteria:

* • Contraindication or refusal to regional anesthesia

  * Contraindication to non-steroidal anti-inflammatory (NSAID's)
  * Allergy to opioids
  * Allergy to paracetamol
  * Creatinine clearance < 30ml/min
  * Weight<50 kg or >100kg
  * Psychiatric disorders and difficulty of communication
  * Lower limb neurological deficit
  * Patients undergoing bilateral or revision total hip replacement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | Day 1
  total morphine dose

SECONDARY OUTCOMES:
pain scores | Hour 2, Hour 4, Hour 6, Hour 12, Hour 18, Hour 24 and on Day 2 and Day 7.
  numerical pain rating scale [1 to 10 worse outcome]
intraoperative opioid consumption | end of surgery
  total fentanyl dose
pain on sitting position | Day 1
  numerical pain rating scale [1 to 10 worse outcome]
QR 9 score | Day 2
  quality of recovery score [0 to 18 best outcome]
ROM | Day 1
  Range of mouvement [0° to 90°best outcome]
pain during walk | Day 7
  numerical pain rating scale [1 to 10 worse outcome]

CONTACTS AND LOCATIONS:
Locations (1):
- Kassab Orthopedic Institute, Manouba, Tunisia

IPD SHARING:
Plan to Share IPD: No